CLINICAL TRIAL: NCT00308477
Title: A Study of the Safety and Efficacy of a New Treatment for Macular Edema Resulting From Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DX4001
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Macular Degeneration; Macular Edema; Branch Retinal Vein Occlusion
Keywords: eye diseases
MeSH Terms: conditions — Macular Degeneration; Macular Edema; Retinal Vein Occlusion; Eye Diseases | interventions — Dexamethasone

INTERVENTIONS:
Drug: dexamethasone

SUMMARY:
This study will evaluate the safety and efficacy of the intravitreal implant of dexamethasone for the treatment of macular edema associated with branch retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Macular edema resulting from branch retinal vein condition
* The criteria for visual acuity and macular thickness are met

Exclusion Criteria:

* History of glaucoma
* Diabetic retinopathy
* Known steroid-responder
* Use of systemic steroids
* Use of Warfarin/Heparin

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Group, Clinical Development Dept., Study Director — Sanwa Kagaku Kenkyusho Co., Ltd.
Locations (12):
- Japan (12):
  - Aichi
  - Chiba
  - Fukuoka
  - Gunma
  - Hokkaido
  - Kagawa
  - Kyoto
  - Mie
  - Miyazaki
  - Osaka
  - Shiga
  - Tokyo